CLINICAL TRIAL: NCT05785533
Title: A Mobile Recovery Guidance App for Children and Young Adults With Acute Ankle Inversion Injuries: a Randomized Controlled Trial
Brief Title: A Mobile Recovery Guidance App for Children and Young Adults With Acute Ankle Inversion Injuries
Acronym: SPRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Naveen Poonai (Other)
Responsible Party: Sponsor-Investigator, Naveen Poonai, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13428
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Ankle Sprains
Keywords: Ankle inversion injury; Mobile app; Recovery guidance
MeSH Terms: conditions — Ankle Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone App (Experimental): The mobile app will allow recording of study outcomes (pain using the vNRS and functional outcomes using the ASKp) and house an interactive educational component to provide daily reminders on pharmacological (ibuprofen and acetaminophen) and non-pharmacological (ice, elevation, and range of motion exercises) for pain management and when to return to activity. The app will collect pain scores using the verbal Numeric Rating Scale (vNRS) and functional outcomes using the Activities Scale for Kids (ASKp) scores on days 3, 5, 7, 10, 12, and 14. The ASKp will be completed by the child with assistance from the caregiver.
  Interventions: Other: Smartphone App
- Standard of Care (Active Comparator): The standard of care group will be asked to read the paper-based discharge instructions in the ED, outlining pharmacological and non-pharmacological pain management and return to activity identical to the information contained in the mobile app. They will download onto their smartphone device a Data Collection App that will only allow them to record the following study outcome measures: daily use of ice, analgesia, range of motion exercises, elevation, and pain using the vNRS and ASKp scores on days 3, 5, 7, 10, 12, and 14. The ASKp will be completed by the child with assistance from the caregiver.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Smartphone App — App that provides recovery guidance based on pain and functional outcomes
  Arms: Smartphone App
Other: Standard of Care — Paper based discharge instruction that provide information on pain management
  Arms: Standard of Care

SUMMARY:
Ankle sprains are the most common musculoskeletal complaint of children presenting to the emergency department (ED). Healing can often be protracted, leading to prolonged pain, missed school and work, and delayed return to a normal activity level. Smartphone apps have been shown to be associated with greater caregiver knowledge and improved outcomes in a number of conditions but have not been explored in ankle sprains. We would like to know if using a smartphone app for children with ankle inversion injuries leads to improved functional outcomes such as pain, mobility, and return to activity. We will be comparing a smartphone app that provides education and daily management reminders to a paper handout to see if the former leads to improved functional recovery.

DETAILED DESCRIPTION:
Acute ankle sprains are one of the most common complaints presenting to primary care offices and EDs. In Canada and the United States, there are more than 2 million ED visits annually due to ankle trauma in children, with 85% of these ankle injuries having no visible bony fracture on radiographs. Furthermore 85% of these ankle sprains are due to forced inversion. Adolescents and young adults have the highest incidence of ankle sprain, with a peak incidence of 7.2 per 1,000 person-years for those 15 to 19 years of age. Although ankle sprains are often perceived as minor injuries, they can have a highly variable prognosis, with up to 64% of patients failing to achieve full recovery and the process may take up to 3 months. Current guidelines are limited in determining prognostic factors associated with functional recovery. The resulting 'one-size fits all' approach to management are controlling acute inflammatory symptoms, using ice and anti-inflammatory medications, alongside early mobilization fails to consider the grade of injury, baseline level of functioning, or individual pain tolerance of the child. Educational guidance individualized to pain beyond the ED may improve functional outcomes.

As of November 2017, 76% of all Canadians own a smartphone, as per Statistics Canada. In a recent study of more than 1600 smartphone phone users in the US, over half (58%) had downloaded a health-related smartphone app. In adult medicine, many health-related smartphone apps have been shown to be associated with greater caregiver knowledge and improved outcomes in allergic rhinitis, post-operative monitoring, and musculoskeletal conditions. In children and adolescents, several studies have explored smartphone apps for asthma and diabetes. To date however, no smartphone apps have been developed for acute musculoskeletal injury management that are directed to children.

This study will examine the utility of a smartphone app to provide discharge instructions and guide treatment using pharmacologic and non-pharmacologic approaches to assist with pain management and return to function in acute ankle inversion injuries, a leading cause of health care visits among children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-30 years
* Presenting to the Paediatric Emergency Department of the Children's Hospital or Adult Emergency Department, London Health Sciences Centre, London, or ntario, St. Joseph Urgent Care Centre, London, Ontario, with a unilateral acute (<= 48 hours) ankle injury based on clinical diagnosis by ED physician
* Able to use a WiFi enabled smartphone with either an iOS or Android operating system with enough memory capability to host the App.

Exclusion Criteria:

* Unable to read or understand English above at least a grade 8 literacy level in the absence of a native language interpreter
* Not independently ambulatory prior to injury (without the use of an assistive device)
* Developmental disability precluding the full comprehension of study-related procedures
* Multi-system or multi-limb injuries
* Concomitant radiographically proven lower extremity fracture or dislocation (with the exception of a suspected Salter-Harris type I injury)

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Activities Scale for Kids - performance version (ASKp) score | Day 7 post-ED discharge
  The ASKp is a self-reported scale of children's physical functioning at home, school, and in the playground. The measure includes 30 questions with total scores ranging from 0 to 100.

SECONDARY OUTCOMES:
Pharmacologic analgesia | Days 1-7 post-ED discharge
  Mean (SD) number of doses of pain medication per day
Non-pharmacologic analgesia | Days 1-7 post-ED discharge
  Mean (SD) number of non-pharmacologic analgesic measures used (ice, elevation) per day
Range of motion (ROM) exercises | Days 1-7 post-ED discharge
  Mean (SD) number of times participant reported performing ROM exercises per day
Verbal Numeric Rating Scale (vNRS) pain score | Day 7 post-ED discharge
  The vNRS is a self-reported pain scale ranging from 0 (no pain) to 10 (maximal pain). The score will reflect the global rating of pain for the day.
Time to return to pre-injury ASKp score | Days 1-14 post-ED discharge
  Number of days until return to pre-injury ASKp score

CONTACTS AND LOCATIONS:
Overall Officials: Janet Knechtel, BA, Study Chair — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Center, London, Ontario, Canada